CLINICAL TRIAL: NCT05474430
Title: Estimating the Risk for and Severity of Respiratory Infections Attributable to CFTR Heterozygosity
Brief Title: Estimating Risk of Respiratory Infections Attributable to CFTR Heterozygosity
Status: Recruiting | Type: Observational
Sponsor: Philip Polgreen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Philip Polgreen, Professor, Internal Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202102125; R01AI143671 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Carrier State; Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasal cells and blood will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Carrier Group: Participants have been identified as Cystic Fibrosis Carriers via previous genetic testing.
- Control Group: Participants have been identified as not being Cystic Fibrosis Carriers via previous genetic testing.

SUMMARY:
A research team member will brush the inferior surface of the subjects' middle turbinate (nasal cavity) using a cytology brush to obtain the cells needed to perform our functional respiratory assays.

An individual trained in phlebotomy will draw one 3 ml lavender top tube of blood to test c-reactive protein, calprotectin, and lactoferrin. They will also draw a 5 ml gold top serum separator tube of blood to test fibroblast growth factor-19.

The participant will answer questions from the baseline survey and report their current medications interview-style with the research team member.

ELIGIBILITY:
CF Carrier Inclusion Criteria:

* Previously tested and shown to be a CF carrier
* English-speaking

Control Group Inclusion Criteria:

* Previously tested and shown to not be a CF carrier or CF patient
* English-speaking

Exclusion Criteria:

* Currently sick with a respiratory infection
* Prisoner Status
* Unable to provide own written, informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CF Carriers and Controls who are not CF carriers.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of Chloride Transport Values | At baseline
  Comparison of chloride transport values in cystic fibrosis carrier group vs control group via t-test.
Comparison of Bicarbonate Transport Values | At baseline
  Comparison of bicarbonate transport values in cystic fibrosis carrier group vs control group via t-test.
Comparison of Airway Surface Liquid pH Values | At baseline
  Comparison of airway surface liquid pH values in cystic fibrosis carrier group vs control group via t-test.
Comparison of Mucous Viscosity Values | At baseline
  Comparison of mucous viscosity values in cystic fibrosis carrier group vs control group via t-test.
Comparison of Bacterial Killing Values | At baseline
  Comparison of bacterial killing values in cystic fibrosis carrier group vs control group via t-test.

SECONDARY OUTCOMES:
Comparison of Fibroblast Growth Factor-19 Values | At baseline
  Comparison of fibroblast growth factor-19 values in cystic fibrosis carrier group vs control group via t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No